CLINICAL TRIAL: NCT05755893
Title: Study of the Unusual Infiltrative Patterns of Malignant Cells and the Immunohistochemical Expression of P53 in Different Histological Types of Endometrial Carcinoma
Brief Title: Unusual Infiltrative Patterns of Malignant Cells in Endometrial Carcinoma and Immunohistochemical Expression of P53
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Adel Adly, principle investigator, Assiut University
Other Study IDs: myometrial invasion, P53
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; tumor budding; microcystic, elongated, fragmented pattern invasion; p53; prognosis
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to clarify the significance of TB, PDC, DR, MELF, and immunohistochemical expression of those infiltrative patterns in patients with endometrial carcinomas (EC). The main questions it aims to answer are:

1. What is the relationship between TB, PDC, DR, MELF, and other clinicopathological features of patients with endometrial carcinomas (EC)?
2. What is the association of TB, PDC, DR, and MELF patterns with disease-free survival and overall survival?
3. Will the evaluation of the immunohistochemical expression of P53 in the TB, PDC, DR, and MELF patterns be important?

DETAILED DESCRIPTION:
Endometrial carcinoma is the most common gynecological tumor in economically developing countries. Because of early symptoms, such as abnormal uterine bleeding, endometrial carcinoma is often diagnosed at an early stage with a favorable prognosis. However, 15-20% of these tumors recur after surgery, leading to poor prognosis.

The International Federation of Gynecology and Obstetrics (FIGO) and the TNM classification are the most widely accepted prognostic classifications. They are based on the assessment of the extent of myometrial invasion and lymph node and distant metastasis. Other tumor characteristics such as histological type and grade, tumor size, and lymphovascular space involvement have also been reported as important prognostic factors. According to risk stratification systems, low-grade and early-stage ECs are classified into low or intermediate-low-risk groups. So, it is necessary to find new parameters to identify patients at a higher risk of relapse among early-stage diagnoses in order to treat and follow them properly without overtreating other patients who remain with an excellent prognosis. This is one of the main gaps that need further improvement in the classification and staging of the disease and this issue needs to be addressed in the near future.

Epithelial-to-mesenchymal transition (EMT), the ability of tumor cells to transform epithelial cell traits into mesenchymal cell traits, is associated with the acquisition of tumor infiltration ability in various carcinomas. Recently, the paracrine signaling of tumor cells and stromal cells in the microenvironment at the tumor invasion front has been shown to play an important role in the induction of EMT. In colorectal cancer, the Wnt/β-catenin signaling pathway that induces EMT is activated in single cells and dedifferentiated tumor cells at the tumor invasion front. Hence, single cells and dedifferentiated tumor cells at the tumor invasion front are believed to be the morphological representations of tumor dedifferentiation and migration associated with EMT. Furthermore, cancer-associated fibroblasts (CAFs) have been reported as a microenvironmental factor related to EMT at the tumor invasion front. CAFs are mobilized by tumor cells via growth factors and cytokines and actively interact with tumor cells in addition to forming a myofibroblastic microenvironment that promotes cancer growth at the tumor invasion front. It has been reported that the paracrine signaling repertoire of tumor cells induces EMT in several cancers.

Single cells, dedifferentiated tumor cells, and CAFs are histopathologically reported as tumor budding (TB), poorly differentiated cluster (PDC), and desmoplastic reaction (DR), respectively in colorectal cancer; each of these is a poor prognostic factor. TB has also been reported as a poor prognostic factor in other carcinomas, including those of the stomach, pancreas, and cervix, and DR has been reported in carcinomas of the pancreas, and thyroid. To our knowledge, TB, PDC, and DR are in EC.

In EC, the microcystic, elongated, and fragmented (MELF) pattern of invasion has been reported as an infiltrative morphology at the tumor invasion front. Therefore, the MELF pattern is also a pathological finding that indicates EMT. Moreover, this pattern has a high frequency of lymphovascular space invasion (LVSI) and lymph node metastasis and occurs in extrauterine disease. By contrast, its effect on long-term prognosis has not been reported and its clinical significance is unclear.

P53 is a Tumor suppressor gene at 17p13, 53 kDa. It ensures that cells repair any damaged DNA before cell division by inducing cell cycle arrest to allow time for DNA repair or to force the cell to undergo apoptosis via activation of the BAX gene Overexpression and complete absence are interpreted as mutation-type, with p53 expression levels in between these extremes are taken as wild type. IHC for p53 protein is available in most pathology labs. This will help us to decide the extent of surgery as complete pelvic and paraaortic node dissection may be considered in endometrial cancers with myometrial invasion having p53 mutation, as it could be detected in about 25% of all endometrial cancer patients .p53 expression pattern was associated with tumor budding status in T1 CRC patients as the rate of p53 positivity was higher in budding tumor compared with tumors without budding.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven Endometrial cancer specimens.
2. underwent total abdominal hysterectomy, with myometrial invasion.

Exclusion Criteria:

1. Endometrial biopsies
2. hysterectomy specimens diagnosed with different pathological lesions rather than EC.
3. Specimens with prior chemotherapy or radiotherapy.
4. specimens without myometrial invasion.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Endometrial cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Unusual infiltrative patterns and their IHC expression P35 | 2 years
  Presence or absence of Tumor budding, microcystic elongated fragmented pattern, desmoplastic reaction and poorly differentiated clusters

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Karamitopoulou E. Role of epithelial-mesenchymal transition in pancreatic ductal adenocarcinoma: is tumor budding the missing link? Front Oncol. 2013 Sep 17;3:221. doi: 10.3389/fonc.2013.00221. PMID 24062980
- [Background] Stewart CJ, Little L. Immunophenotypic features of MELF pattern invasion in endometrial adenocarcinoma: evidence for epithelial-mesenchymal transition. Histopathology. 2009 Jul;55(1):91-101. doi: 10.1111/j.1365-2559.2009.03327.x. PMID 19614771
- [Background] Park JY, Hong DG, Chong GO, Park JY. Tumor Budding is a Valuable Diagnostic Parameter in Prediction of Disease Progression of Endometrial Endometrioid Carcinoma. Pathol Oncol Res. 2019 Apr;25(2):723-730. doi: 10.1007/s12253-018-0554-x. Epub 2019 Jan 2. PMID 30604272
- [Background] Kobel M, Ronnett BM, Singh N, Soslow RA, Gilks CB, McCluggage WG. Interpretation of P53 Immunohistochemistry in Endometrial Carcinomas: Toward Increased Reproducibility. Int J Gynecol Pathol. 2019 Jan;38 Suppl 1(Iss 1 Suppl 1):S123-S131. doi: 10.1097/PGP.0000000000000488. PMID 29517499
- [Background] Yamamoto M, Kaizaki Y, Kogami A, Hara T, Sakai Y, Tsuchida T. Prognostic significance of tumor budding, poorly differentiated cluster, and desmoplastic reaction in endometrioid endometrial carcinomas. J Obstet Gynaecol Res. 2021 Nov;47(11):3958-3967. doi: 10.1111/jog.14997. Epub 2021 Aug 26. PMID 34448279